CLINICAL TRIAL: NCT02647216
Title: Mindfulness Training to Improve Well-being in Post-Treatment Breast Cancer Patients
Brief Title: Mindfulness for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14-01138
Record Dates: First submitted 2015-12-30; First posted 2016-01-06 (Estimated); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Anxiety; Depression; Breast Cancer
Keywords: Mindfulness Based Cognitive Therapy (MBCT); anxiety; depression
MeSH Terms: conditions — Anxiety Disorders; Depression; Breast Neoplasms | interventions — Mindfulness-Based Cognitive Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Based Cognitive Therapy (MBCT) (Active Comparator): MBCT is a structured 8-week group intervention which integrates aspects of cognitive behavioral therapy (CBT) with components of the Mindfulness Based Stress Reduction (MBSR) program.
  Interventions: Behavioral: Mindfulness Based Cognitive Therapy
- Treatment as Usual (TAU) (Active Comparator): Subjects randomized to TAU will be advised to seek help from their family doctor or other sources as they normally would if they encountered symptomatic deterioration or other difficulties over the course of the study. All treatments received over the course of the study (for the TAU group) and outside of the study (for the MBCT group) will be assessed at the 3-month follow up (Visit 3).
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Mindfulness Based Cognitive Therapy — Weekly MBCT sessions consist of: a) mindfulness practice including breath-focused sitting meditation, body scanning, and mindful stretching; b) review of previous weeks' homework and an overview of the current week's homework; c) barriers to completing the homework. Homework includes: a) practicing the mindfulness exercise reviewed in class using the CDs provided to each participant (guided practice of the relevant exercise); b) maintaining a calendar of pleasant events; c) mindfully engaging in activities of daily living; and d) logging practice efforts in a daily log.
  Arms: Mindfulness Based Cognitive Therapy (MBCT)
Behavioral: Treatment as Usual — Subjects randomized to the Treatment as Usual group will be advised to seek help from their family doctor or other sources as they normally would if they encountered symptomatic deterioration or other difficulties over the course of the study.
  Arms: Treatment as Usual (TAU)

SUMMARY:
The primary purpose of this study is to evaluate the effects of Mindfulness Based Cognitive Therapy (MBCT) vs. Treatment as Usual (TAU) for depression and anxiety symptoms in breast cancer patients in recovery. Investigators will examine whether MBCT-related improvements in sleep quality, illness-related distress, and rumination (escalating cycles of negative thinking) predict MBCT-related decreases in depression and anxiety symptoms (Aim 2). Exploratory analyses will examine whether demographics (e.g., age, sex, race/ethnicity), individual differences (e.g., perceived stress, social support), clinical characteristics (e.g., stage/severity of diagnosis), and treatment adherence (e.g., sessions attended, hours of weekly practice) help determine for whom MBCT is most effective (Aim 3).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over
* Able to speak and read English
* Diagnosis of breast cancer (any stage) for which active treatment (e.g., surgery, chemotherapy, and/or radiotherapy) has been completed within 2 months to 2 years

Exclusion Criteria:

* Cognitive impairment or mental illness that would impair ability to provide consent or participate in the program;
* Major psychiatric disorder (e.g., psychosis, personality disorder)
* Current suicidal ideation or suicide attempt within past 3 months
* Past participation in an MBCT group

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Change in Anxiety Level using the State-Trait Anxiety Inventory (STAI)-Form Y | 3 Months
  This measure consists of 20-items that assess trait anxiety and 20 for state anxiety.
Change in level of Depression using the Beck Depression Inventory-II (BDI-II) | 3 Months
  The 21-item version of this widely used measure will be used to assess depressive symptoms.

SECONDARY OUTCOMES:
Change in Quality of Life using the Patient Reported Outcomes Measurement Information System (PROMISE) | 3 Months
  PROMISE: 10 Item measure of quality of life
Change in fatigues score using a Functional Assessment of Cancer Therapy Breast and Fatigue subscales (FACIT-B and F): | 3 Months
Change in Physical Health Symptoms | 3 Months
Change in Sleep Quality using the Pittsburgh Sleep Quality Index (PSQI): | 3 Months
  This 19-item measure assesses habitual sleep quality over the last month. It consists of 7 subscales (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, daytime dysfunction), and also provides a global sleep quality score.
Change in Illness Perceptions using the Brief Illness Perception Questionnaire (B-IPQ) | 3 Months
Change in Rumination using the Ruminative Responses Scale (RSS): | 3 Months
  Change in the level of escalating cycles of negative thinking

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Spruill, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States